CLINICAL TRIAL: NCT06815016
Title: The Effect of Adding Reflexology to Mulligan Mobilization for Patient With Knee Osteoarthritis
Brief Title: Reflexology and Mulligan Mobilization for Knee Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rania Ahmed Nassar, demonstrator physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005479
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Knee Osteoarthritis; Knee Osteoarthritis (Knee OA)
Keywords: Knee Osteoarthristis; reflexology; Mulligan's Mobilization
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Congresses as Topic; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Reflexology and conventional (Experimental): treatment all patient with knee osteoarthritis three times per week
  Interventions: Other: reflexology and conventional
- mulligan mobilization and conventional (Experimental): treatment all patient with knee osteoarthritis three times per week
  Interventions: Other: mulligan mobilization and conventional
- Reflexology ,mulligan mobilization and conventional (Experimental): treatment all patient with knee osteoarthritis three times per week
  Interventions: Other: Reflexology ,mulligan mobilization and conventional; Other: mulligan mobilization and conventional
- Conventional methods (Experimental): treatment all patient with knee osteoarthritis three times per week
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Reflexology ,mulligan mobilization and conventional — Reflexology is a systematic practice in which applying some pressure to any particular points on the feet and hands give impacts on the health of related parts of the body as (Knee reflex point, Pituitary reflex point, Entire spine, Liver reflex area, Thyroid reflex area ) Mulligan's Mobilization with Movement (MWM) apply accessory gliding force combined with active movement as (Lateral glide MWM for flexion / extension, Medial glide MWM for flexion / extension, Self-medial glide MWM for knee flexion/extension: home exercise)
  Arms: Reflexology ,mulligan mobilization and conventional
Other: reflexology and conventional — Reflexology as (Knee reflex point, Pituitary reflex point, Entire spine, Liver reflex area, Thyroid reflex area ) and conventional methods as (Transcutaneous Electrical Nerve Stimulation (TENS), Ultrasound Therapy and exercises) treatment.
  Arms: Reflexology and conventional
Other: mulligan mobilization and conventional — Mulligan mobilization as (Lateral glide MWM for flexion / extension, Medial glide MWM for flexion / extension, Self-medial glide MWM for knee flexion/extension: home exercise) and conventional methods as (Transcutaneous Electrical Nerve Stimulation (TENS), Ultrasound Therapy and exercises) treatment.
  Arms: Reflexology ,mulligan mobilization and conventional; mulligan mobilization and conventional
Other: Conventional treatment — Conventional methods as (Transcutaneous Electrical Nerve Stimulation (TENS), Ultrasound Therapy and exercises) treatment.
  Arms: Conventional methods

SUMMARY:
to investigate the effect of adding Reflexlogy to mulligan mobilization and the conventional treatment for patients with Osteoarthritis knees

DETAILED DESCRIPTION:
Knee osteoarthritis (OA), also known as degenerative joint disease, is typically the result of wear and tear and progressive loss of articular cartilage. Treatment by reflexology stimulation increases blood flow to the associated organ or body part. On the other hand, the nerve impulse theory claims that reflexology stimulation boosts nervous connection to the conforming body parts. Regarding to the energy theory; organs and body parts are connected through electromagnetic fields and that these pathways are blocked in states of disease. Finally, lactic acid theory pointed that lactic acid accumulates on the soles of the feet in the form of crystals which promotes free circulation, so reduces regular flow .The effects of foot reflexology on improving physical complains of KOA. Therefore, this study was conducted to evaluate the effectiveness of reflexology foot massage on pain intensity and physical functional abilities among patients with Knee Osteoarthritis.

Mulligan's Mobilization with Movement (MWM) advocates therapist-applied accessory gliding force combined with active movement The goal of MWM is to achieve immediate pain relief possibly by regulation of the non-opioid pain sensory pathways and by correction of micro positional faults. These positional faults may result from changes in the shape of articular surfaces, cartilage thickness, fiber orientation in the capsule-ligamentous complex, and the direction of musculo-tendinous pull, causing altered mechanics in the osteoarthritic knees.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 40 years.
2. Body Mass Index ≤30 kg/m².
3. All participants have Calcium Deficiency
4. Osteoarthritis in mild and moderate stage not in the acute stage
5. The subjects were chosen from both genders

Exclusion Criteria:

1. Deep Vein Thrombosis
2. Fractures
3. Gangrena Patient
4. Osteopenic Patient
5. Lactating or pregnant women
6. Cancer
7. Neurological conditions.
8. Patients with injury including; (lesions, sprain, open wounds, foot ulcer and or burn of the lower extremities), hemorrhage, epilepsy, irregular heartbeat.
9. Vascular (Anticoagulant Therapy, Aortic Aneurysm)
10. Neurological Deficits (multilevel PIVD, Cervical Myelopathy)
11. Psychological Disorders.

    -

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale | one month
  consists of a line, usually 10 cm long, ranging from no pain or discomfort (zero), to the worst pain that could possibly feel (10)

SECONDARY OUTCOMES:
The Knee Injury and Osteoarthritis Outcome Score (KOOS) | one month
  The Knee injury and Osteoarthritis Outcome Score (KOOS) was developed as an extension of the WOMAC Osteoarthritis Index with the purpose of evaluating short-term and long-term symptoms and function in subjects with knee injury and osteoarthritis. The KOOS holds five separately scored subscales: Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL)

OTHER OUTCOMES:
Kinovea | one month
  Kinovea is a free software that uses a virtual goniometer to measure joints for measure Flexion and Extension ROM of knee

CONTACTS AND LOCATIONS:
Overall Officials: Noran A Elbehary, Professor of physical Therapy, Principal Investigator — basic science department, faculty of physical therapy cairo university; Mariam O Grase, lecturer physical therapy, Principal Investigator — basic science department, faculty of physical therapy cairo university
Locations (1):
- Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Bakir E, Baglama SS. The Effect of Foot Reflexology and Knee Massage With Black Cumin Seed Oil on Knee Osteoarthritis Symptoms. Holist Nurs Pract. 2026 Jan-Feb 01;40(1):56-65. doi: 10.1097/HNP.0000000000000714. Epub 2025 Nov 11. PMID 39642267
- [Background] Bhagat M, Neelapala YVR, Gangavelli R. Immediate effects of Mulligan's techniques on pain and functional mobility in individuals with knee osteoarthritis: A randomized control trial. Physiother Res Int. 2020 Jan;25(1):e1812. doi: 10.1002/pri.1812. Epub 2019 Sep 10. PMID 31502354